CLINICAL TRIAL: NCT07306780
Title: Barriers to Dental Care: Exploring the Role of Procrastination in Seeking Care
Brief Title: Procrastination in Seeking Dental Care
Status: Enrolling by invitation | Type: Observational
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Other Study IDs: Navi Bansal
Record Dates: First submitted 2025-12-02; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Procrastination

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Irrational Procrastination Scale (IPS) — Irrational Procrastination Scale is a 9-item questionnaire to assess one's level of procrastination. Respondents rate how often each statement is true of them on a 5-point scale. Items 2, 5, and 8 are reverse scored. Higher total scores indicate greater tendencies toward procrastination
Other: Oral Health Self Efficacy Scale (OHSES) — An Oral Health Self-Efficacy Scale (OHSES) is a tool used to measure a person's confidence in their ability to maintain good oral health. Participants rate their confidence on a scale, for example, from "Not at all confident" to "Strongly confident" or "Strongly disagree" to "Strongly agree". Responses are summed to get a total score, with a higher score indicating greater self-efficacy in oral health.

SUMMARY:
Patients fulfilling the eligibility criteria will be enrolled in the study will be given online survey to fill questionnaire.

Questionnaire will be provided to the patient which include the questions about following parameters:

1. Socio-Demographic factors
2. Self-reported oral health and dental satisfaction
3. Dental attendance regarding regular, past and future dental visits.
4. Delay of dental care Procrastination will be measured using Irrational Procrastination Scale (IPS). Self-Efficacy for oral Health will be measured using Oral Health Self-Efficacy Scale (OHSES)

ELIGIBILITY:
Inclusion Criteria:• Individuals who were able to read and understand English language.

* Individuals who were above the age of 18 years and consented to participate in the study.

Exclusion Criteria: Patients who were unwilling to take part in the study.

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants with age above 18 years will be recruited in the study. Recruitment of the patients for the study will be based on eligibility criteria after obtaining informed consent.
Sampling Method: Probability Sample
Enrollment: 196 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Effect of Procrastination on Dental Attendance | Day 1
  Correlation coefficient between Irrational Procrastination Scale (IPS) score and dental attendance. IPS scale is a 9-item scale where participants respond to a statement on a Likert scale from 1 to 5 in order to indicate whether the statement describes them well (5) or not (1). Score range 9-45
Effect of Oral Health Self Efficacy on dental attendance | Day 1
  Correlation coefficient between Oral health self efficacy scale (OHSES) score and dental attendance. OHSES is a 12-item scale to which respondents agreed or disagreed on a Likert scale (1-5). Score range 12-60

CONTACTS AND LOCATIONS:
Locations (1):
- PGIDS Rohtak, Rohtak, Haryana, India